CLINICAL TRIAL: NCT03681587
Title: How to Give Back the Pleasure of Eating to the Dependent elderly_observational Study
Brief Title: How to Give Back the Pleasure of Eating to the Dependent Elderly
Acronym: Petit-dejeuner
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VVW 2017 Petit-dejeuner
Record Dates: First submitted 2018-08-27; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Elderly People; Breakfast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Control situation — Standard breakfast usually offered "monotonous control condition" at the retirement home: the time of distribution, the duration of ingestion and the composition will be habitual. This meal and subsequent meals will be measured over 3 consecutive days with observation periods at breakfast time in order to identify the variables of pleasure, feasibility, commensality and conviviality in 2 situations: alone in the room or with others in the dining room.
Other: Experimental situation — Salty/sweet breakfast "varied experimental situation": the time of distribution and the duration of mealtime will be open and the composition will be varied with sweet/savory foods. This meal and subsequent meals will be measured over 3 consecutive days with observation periods at breakfast time in order to identify the variables of pleasure, feasibility, commensality and conviviality in 2 situations: alone or in the room or with others in the dining room.

SUMMARY:
Many public health recommendations and policies aim to combat malnutrition in the elderly. It must be noted that levels of malnutrition are high in the elderly with more than 70% of the dependent population at home or in institutions and 30 to 70% of elderly people in hospitals.

In hospitals, the collective catering system and the "medicalisation" of meals (diets, medicines, etc.) force patients to change their eating habits, and they are often faced with a lack of choice and a less pleasurable experience. These organizational constraints are particularly harmful for elderly patients who tend to be malnourished or at risk of malnutrition and who are often polypathological and polymedicated.

If eating is one of the only pleasures sometimes left to this fragile population, breakfast is one of the most appreciated meals of the day (after a fasting time >10h). It tends to follow the habits acquired at home and is mostly oriented towards sweet foods. However, it is not known whether different and more varied choices could change dietary directions and intakes.

Offering sweet and savoury foods can upset medical prescriptions, cultural habits and can go against what remains a patient need: the pleasure of eating.

Although some work in the medico-social field has been successfully carried out and has reported changes in dietary behaviour in a choice situation (buffet type) at breakfast, scientific studies have not yet been done in a retirement home environment. The objective of this project is to emphasize the sensory pleasure and commensality of breakfast. During this buffet meal, sweet and savoury foods will be offered. The idea is to detect if the variety will naturally direct individual choices towards the savory and/or sweet flavours and if it encourages an increase in caloric and protein intakes. Several studies have shown that sensory changes in the elderly can lead to changes in behaviour and food preferences. The decrease in the pleasure only accentuates the causes of malnutrition. Moreover, preconceived ideas reinforce the association between the elderly and a preference for sweet foods. However, no study has shown that the elderly find less pleasure in savory than sweet foods, especially at breakfast.

The research will be organized as follows:

Phase 1: follow-up of breakfast consumption by food weighing. This is a prospective study that will be carried out at Dijon University Hospital within the retirement home.

The consumption of each meal will be measured the day of the breakfast with savory and sweet options, and then two days after in usual conditions in the individual's room. The distribution, service and consumption methods will be consistent with the habits of the units where the investigation is taking place.

For each resident, food consumption will be recorded three times, at one month intervals over 2 non-consecutive days.

Phase 2: observations at breakfast time Pleasure evaluation - Feasibility - commensality - conviviality A SWOT (Strengths, Weaknesses, Opportunities and Threats) analysis will be conducted for each type of environment and meals offered. This analysis will be done using established grids and semi-directive interviews with resource persons who are working in the field (the professionals involved), and with research support units. The professionals will be asked to complete various scales, of the Likert type, before and after the breakfasts included in the study.

ELIGIBILITY:
Inclusion Criteria:

* persons over 75 years of age
* person residing in a retirement home
* orally fed person
* person who speaks and understands French

Exclusion Criteria:

* person not affiliated to a social security scheme
* person requiring enteral or parenteral feeding
* dying person

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly people residing in a retirement home
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of Ingesta weight at 2 months | Month 0, 1 and 2

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France